CLINICAL TRIAL: NCT01805375
Title: A Cancer Research UK Phase I Trial of the Anti-CD19 DI-B4 Monoclonal Antibody Given Intravenously, Weekly for Four Weeks, in Patients With Advanced CD19 Positive Indolent B-cell Malignancies
Brief Title: A Phase I Trial of DI-B4 in Patients With Advanced CD19 Positive Indolent B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CRUKD/12/003
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Indolent B-cell Lymphoma; Chronic Lymphocytic Leukaemia; Waldenström Macroglobulinaemia
Keywords: Phase I, Cancer, CD19 positive, B-Cell lymphoma, chronic lymphocytic leukaemia; Waldenström Macroglobulinaemia
MeSH Terms: conditions — Leukemia, B-Cell; Waldenstrom Macroglobulinemia; Neoplasms; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: DI-B4 — DI-B4 will be administered once weekly for up to a total of four weeks. The starting dose will be 0.02 mg given as an intravenous infusion. A cycle is 1 week in duration and patients should expect to receive a maximum of 4 cycles.

SUMMARY:
The main aims of this clinical study are to find out the maximum dose that can be given safely to patients, the potential side effects of the drug and how they can be managed. The study will also look at what happens to Anti-CD19 (DI-B4) inside the body.

DI-B4 is a type of drug called an Anti-CD19 monoclonal antibody which is being used to stop the growth and kill cancerous immune cells by targeting the B-cell marker (CD-19) expressed on their surface. This drug has not been given to patients before.

DI-B4 will be given weekly by intravenous infusion for four weeks. The study is in two parts. In Part 1, small groups of patients will be treated at increasing doses to find the highest safest dose and best dose for part 2 of the study. Approximately 16-20 patients will be treated in this part. In Part 2, the dose identified in Part 1 will be given to approximately 20 patients.

Patients recruited to the study will receive four weeks (cycles) of treatment. They will attend an end of therapy visit eight weeks after their last dose of DI-B4, and attend follow-up visits up to eighteen months after their first dose of DI-B4. Information on the overall and progression free survival will be collected for a period up to eighteen months after the final patient is treated on the study.

Patients will have blood and urine samples taken each week during treatment amongst other clinical tests. CT scans will be performed at the start of the study, at eight weeks post treatment and six months after the study start. Bone marrow biopsies and FDG-PET scans will only be taken if needed. Research blood samples will also be taken to look at what happens to the drug inside the body.

It is important to explain that patients will have advanced cancer so it is unlikely that patients will benefit directly from taking part but the study may help improve future treatment of cancer.

DETAILED DESCRIPTION:
Patients with relapsed or refractory CD19 positive indolent B-cell lymphoma, Waldenström Macroglobulinaemia or chronic lymphocytic leukaemia will be entered into this study.

For the vast majority of patients, B-cell non Hodgkin lymphoma and chronic lymphocytic leukaemia are incurable using existing therapeutic approaches.

Although anti-CD20 directed therapy has improved outcomes, more than fifty percent of patients still relapse following treatment or are refractory to it and therefore additional novel non-cross resistant therapies are urgently required.

DI-B4 is a humanised, low-fucosylated anti-CD19 Immunoglobulin (Ig) G1 monoclonal antibody with potent antibody-dependent cell-mediated cytotoxicity (ADCC) but minimal complement dependent cytotoxicity (CDC). The target antigen, CD19, is the canonical B-cell marker that is expressed on all B-cells including the malignant B-cells in NHL, CLL and acute lymphoblastic leukaemia (ALL). The CD19 antigen is therefore an attractive B-cell lineage specific target for monoclonal antibody therapy. DI-B4 is expected to act through the depletion of normal and malignant CD19 positive cells, primarily via ADCC.

This is a multi-centre, Phase I, dose escalation/dose expansion study. For the first three cohorts, an intra-patient dose escalation scheme will be followed unless a DLT is observed. From Cohort 4 onwards, a standard 3 + 3 dose escalation schedule of DI-B4 will be continued until the maximum tolerated dose (MTD) is defined, up to a maximum dose of 1000mg.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven relapsed or refractory indolent B-cell lymphoma or chronic lymphocytic leukaemia. Patients must have received at least one line of previous therapy.

2. CD19 positive malignancy as demonstrated by immunohistochemistry or flow cytometry

3. Life expectancy of at least 12 weeks

4. World Health Organisation (WHO) performance status of 0-1

5. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient commences treatment with DI-B4.

Laboratory Test Value required Haemoglobin (Hb) ≥ 9.0 g/dL (red cell support is permissible), Absolute neutrophil count (ANC) ≥1.0 x 10^9/L (or ≥0.5 x 10^9/L if bone marrow involvement), Platelet count ≥75 x 10^9/L (or ≥30 x 10^9/L if bone marrow involvement), Serum bilirubin ≤1.5 x upper limit of normal (ULN), unless raised due to Gilbert's syndrome in which case up to 3 x ULN is permissible Alanine amino-transferase (ALT) and/or aspartate amino-transferase (AST) ≤ 2.5 x (ULN) unless raised due to hepatic involvement in which case up to 5 x ULN is permissible

6. 18 years or over

7. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

8. Indolent B-cell lymphoma patients only: Patient has either at least one measurable lesion by CT scan (defined as >1.5 cm in one axis) or in the case of Waldenström's macroglobulinemia, disease must be assessable by the protocol criteria.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, chemotherapy or investigational medicinal products during the previous 4 weeks before treatment.

2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Drug Development Office (DDO) should not exclude the patient.

3. Known to be serologically positive for hepatitis B (unless due to vaccination), hepatitis C or human immunodeficiency virus (HIV).

4. Patients with clinically active leptomeningeal or central nervous system lymphoma/leukaemia.

5. Patients with transformed lymphoma from a pre-existing indolent lymphoma. Patients with a previous history of transformation, but on this disease episode have a biopsy proven indolent recurrence may be included.

6. Patients receiving corticosteroids, except where the patient has been on a stable dose for the preceding seven days. Doses of prednisolone or equivalent >10 mg daily are not permitted whilst on the study, doses up to 20mg can be taken any time prior to Cycle 1, Day 1

7. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), history of unstable angina pectoris or myocardial infarction up to 1 year prior to patient enrolment into the trial, presence of severe valvular heart disease or presence of a ventricular arrhythmia requiring treatment

8. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) during the trial and for six months afterwards are considered eligible.

9. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

10. Major thoracic or abdominal surgery from which the patient has not yet recovered.

11. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.

12. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of DI-B4. Participation in an observational trial would be acceptable.

13. Any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
To recommend a dose for future trials with a new drug called DI-B4 by finding the highest safe dose which can be given to patients | 38 Months

SECONDARY OUTCOMES:
Measuring of PK parameter values for DI-B4 including AUC, Cmax, Tmax, and half life T1/2. | Samples taken during the four weeks of treatment and analysed in batches per cohort within 6 months of sampling
To evaluate the effect of DI-B4 on the depletion of peripheral blood and bone marrow B-cells. | Samples taken during the four weeks of treatment, and for 18 month follow-up and analysed in batches per cohort within 6 months of sampling
To look for signs of anti-tumour activity of DI-B4 in patients with relapsed or refractory indolent B-cell malignancies. | 38 months
To assess immunogenicity of DI-B4 in patients with relapsed or refractory indolent B-cell malignancies | 54 months
To measure the time to disease progression and eighteen month survival | 54 months

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Royal Liverpool and Broadgreen University Hospital NHS Trust, Liverpool
  - The Christie NHS Foundation Trust, Manchester
  - The Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton